CLINICAL TRIAL: NCT06720636
Title: Ultralong-segment Barrett's Esophagus: Towards a Capsule-sponge Surveillance Strategy
Acronym: ULSBE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Cyted Health Inc (Industry); University of Cambridge (Other)
Responsible Party: Principal Investigator, Judith Honing, Principal Investigator, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL87577.078.24
Record Dates: First submitted 2024-11-21; First posted 2024-12-06 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Barrett Esophagus
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study group (Experimental): Subjects will receive the EndoSign test prior to their scheduled clinically indicated upper endoscopy by an expert endoscopist, per routine standard of care. Additional biopsies will be taken and 10cc of blood will be collected from the cannula used for sedation. Subjects will also receive three questionnaires regarding baseline characteristics, gastrointestinal symptoms and acceptability.
  Interventions: Device: EndoSign

INTERVENTIONS:
Device: EndoSign — The EndoSign cell collection device is a non-endoscopic capsule sponge device used to collect pan-esophageal samples.
  The Endosign procedure consists of an expandable, spherical mesh, which is attached to a string and contained within a soluble capsule. Seven minutes after swallowing (once the capsule has dissolved), the spherical mesh, which measures around 3cm in diameter is retrieved by pulling on the string. Upon retrieval the capsule-sponge scrapes against the surface of the top of the stomach and esophagus and collects epithelial cells. The capsule-sponge sample is then placed into a preservative fluid and the specimen is processed for molecular tests.

SUMMARY:
The purpose of this study is to evaluate the Endosign capsule sponge test as a novel surveillance method in patients with an ultralong-segment Barrett's esophagus.

DETAILED DESCRIPTION:
In this study we will investigate the concordance between the Endosign capsule sponge test and esophagogastroduodenoscopy (EGD) by an expert endoscopist to detect dysplasia and/or esophageal adenocarcinoma (EAC) in patients with an ultralong-segment Barrett's esophagus. Patients will receive both the Endosign test and an EGD, after which we will compare both outcomes. To detect dysplasia and/or EAC on the cells collected by the Endosign test, we will look at cellular atypia and use p53 immunohistochemistry and novel biomarkers. In the future the Endosign test could perhaps replace EGD in the surveillance of Barrett's esophagus patients.

ELIGIBILITY:
Inclusion Criteria:

* Any participant 18 years and above, with ultralong-segment Barrett's esophagus and clinically fit for an endoscopy
* Ability to provide informed consent

Exclusion Criteria:

* Individuals with a diagnosis of an oro-pharynx, esophageal or gastro-esophageal tumor (T2 staging and above), or symptoms of dysphagia
* Esophageal varices or stricture requiring dilatation of the esophagus
* Individuals who have had a cerebrovascular event < 6 months prior where their swallowing has been affected
* Patients who have had previous treatments such as Photodynamic therapy (PDT), Radiofrequency ablation (RFA) or Argon Plasma Coagulation (APC) for dysplastic Barrett's esophagus
* Participants who are unable to provide informed consent
* Participants under age 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Concordance between EndoSign and upper endoscopy to detect dysplasia and/or esophageal adenocarcinoma | 3 years
  We will determine the concordance between the EndoSign test and upper endoscopy by an expert endoscopist to detect dysplasia and/or esophageal adenocarcinoma in patients with an ultralong-segment Barrett's esophagus.

SECONDARY OUTCOMES:
Patient rating of both the EndoSign procedure and upper endoscopy on an experience scale | 3 years
  Patients with an ultralong Barrett esophagus will rate their experience with both the Endosign procedure and endoscopy on a scale from 1 - 10, with 1 being the worst experience ever and 10 the best experience ever. These results will be compared to assess which procedure is generally more acceptable to patients.
Sensitivity & specificity | 3 years
  To determine the sensitivity and specificity of the EndoSign to detect any form of dysplasia or esophageal adenocarcinoma in a cohort of ultralong-segment Barrett's esophagus patients.
Additional value of p53 immunohistochemistry | 3 years
  To determine the additional value of p53 immunohistochemistry in risk stratifying patients with ultralong-segment Barrett's esophagus.
Accuracy of a new risk stratification model for neoplastic progression | 3 years
  We will determine the accuracy of a newly developed risk stratification model that predicts which patients with an ultralong-segment Barrett's esophagus have the highest chance of neoplastic progression. We will use both clinical risk factors and p53 immunohistochemistry.
Accuracy of a new shallow Whole Genome Sequencing assay to predict neoplastic progression | 3 years
  We will determine the accuracy of a new shallow Whole Genome Sequencing (sWGS) assay for predicting neoplastic progression in patients with an ultralong Barrett's esophagus.
Validation of the sensitivity of a current methylation-based sequencing approach to predict neoplastic progression | 3 years
  We aim to validate the sensitivity of a current sequencing approach using both methylation and genome instability to detect neoplastic progression in patients with an ultralong Barrett's esophagus.

CONTACTS AND LOCATIONS:
Overall Officials: Judith Honing, MSc, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus Medisch Centrum, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No